CLINICAL TRIAL: NCT04710147
Title: Cross-cultural Adaptation to the Spanish Population and Validation of Community Balance & Mobility Scale in Persons With Acquired Brain Injury in Subacute and Chronic Phase
Brief Title: Cross-cultural Adaptation to the Spanish Population and Validation of the Community Balance & Mobility Scale (S-CB&M)
Acronym: S-CB&M
Status: Completed | Type: Observational
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Centro de Referencia Estatal de Atención Al Daño Cerebral (Other)
Responsible Party: Principal Investigator, Cristina Lirio, Principal Investigator, University of Castilla-La Mancha
Other Study IDs: CLirio05
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Brain Injury, Chronic
Keywords: Acquired Brain Injury; Balance Assessment; Central Nervous System Diseases
MeSH Terms: conditions — Brain Injury, Chronic; Brain Injuries; Central Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to acquired brain injury (ABI), is often difficulty in gait and balance alterations, as problems that patients designated as the most disabling. It is essential to an effective assessment of the balance.

Objective: The purpose of the present project adapt and verify the validity of the scale Community Balance and Mobility (CB&M), in patients with ABI in subacute and chronic stage, since that is postulated as a brief tool and covering the peculiarities of the specific alterations of the patient after suffering brain injury.

Methodology: Between February 2021 and June 2022 will be transcultural adaptation to the ABI population and validation of psychometric scale CB&M in three phases. 100 subjects who receive treatment in centers of attention to brain injury in Spain will be recruited.

Results: validity and reliability parameters shall be calculated by means of descriptive statistics for each item of the scales and the set of scale score. Investigators will also analyze the internal consistency using Cronbach's alpha, the interclass correlation coefficient will be used to determine the reliability, and the items will be scanned with the Pearson coefficient: > 0.20, among other parameters.

DETAILED DESCRIPTION:
Cristina Lirio-Romero et al., will develop a cross-cultural adaptation to the Spanish population with Acquired Brain Injury (ABI) and psychometric validation of the Community Balance and Mobility (CB&M) scale. The author of the scale has consented the adaptation of the scale. The study will take place at several centers of attention to brain injury in Spain. After receiving the approval of the Ethics and Clinical Research Committee of the University of Alcalá (Madrid), it is proposed to implement the study between February 2021 and June 2022. A minimum of 100 adults, aged between 18 and 65, will be recruited subacute or chronic state after suffering brain injury. The sample size conforms to COSMIN recommendations.

After verifying that there are no parallel studies on the subject in progress, the possible participants will be informed of the development of the investigation (ANNEX 1), who must sign the informed consent (ANNEX 2) before being recruited into the study. In addition, a coding sheet (ANNEX 3) of the participants will be filled in so that from now on the data related to the proper name does not appear but with a number that ensures the protection of their data.

Selection criteria to enter to participate in the study will be: adults who had suffered a ABI at least 2 months ago, that their disability before suffering it was less than or equal to three on the scale modified by Rankin, who have an absence of cognitive impairment according to the Minimental State Examination scale, that is, a score in it greater than 24, without previous diseases that alter the balance, that were clinically stable and without fever, with the ability to walk with help technical or without it, and that they gave their informed consent.

On the other hand, those people with medical contraindications for physical tests (acute musculoskeletal or peripheral nervous system disorders), who did not understand the instructions, severe aphasias or with subjects with acute processes of any added pathology will be excluded.

The study was developed in 3 phases:

Phase 1: Transcultural adaptation process. Phase 2: Pre-Test: collected , as well as the ease of interpretation of the results.

Phase 3: Psychometric validation process.

ELIGIBILITY:
Inclusion Criteria:

* The participants will be users from centers of attention to brain injury.
* Adults who had suffered a ABI, at least 2 months before.
* The disability before suffering ABI was less than or equal to three on the scale modified Rankin.
* Lack of cognitive impairment scale Minimental State Examination, with a score is > 24.
* No previous diseases that alter the balance.
* Clinically stable and without fever-
* Ability to walk with technical support or without it.
* Signing an informed consent.

Exclusion Criteria:

* Medical contraindications to perform physical tests (acute or peripheral nervous system musculoskeletal disorders).
* Not understand the instructions.
* Subjects with severe aphasia.
* Subjects with acute processes of any added pathology.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spanish population with Acquired Brain Injury.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
1. Test-retest Reliability | 2 months
  the overall consistency measures the homogeneity of the scale and the interdependence of the items, indicating the relationship between them.
  To determine test-retest test reliability, the intraclass correlation coefficient (ICC) will be used. Derived from the test-retest reliability study, the measurement error will be calculated, using the formula standard deviation (SD) x √1-ICC.
Validity | 2 months
  To analyze the convergent validity, it will be applied on the first day of the week and before receiving treatment.
Berg Balance Scale | 2 months
  It evaluates deficiencies in balance in response to 14 points ranging from 0-worst balance to 4-best balance (total 56 points). Berg Balance Scale is the gold standard of comparison for obtaining validity

SECONDARY OUTCOMES:
Sensitivity to change | 2 months
  Ability of Community Balance and Movility to detect real changes in the health of the subjects, whether positive or negative (from 0-worse to 96-better balance and mobility).
  The differences in the scores between the periods of the beginning of any proposed treatment and at the end of this will be evaluated by the effect size and the standardized response to the change.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Lirio-Romero, PhD, Principal Investigator — University of Castilla-La Mancha; Marta Fernández-Hontoria, BsC, Study Chair — Centro de Referencia Estatal de Atención Al Daño Cerebral
Locations (1):
- Cristina Lirio-Romero, Toledo, Spain

REFERENCES:
- [Background] Perennou D, Decavel P, Manckoundia P, Penven Y, Mourey F, Launay F, Pfitzenmeyer P, Casillas JM. [Evaluation of balance in neurologic and geriatric disorders]. Ann Readapt Med Phys. 2005 Jul;48(6):317-35. doi: 10.1016/j.annrmp.2005.04.009. French. PMID 15932776
- [Background] Wild D, Grove A, Martin M, Eremenco S, McElroy S, Verjee-Lorenz A, Erikson P; ISPOR Task Force for Translation and Cultural Adaptation. Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes (PRO) Measures: report of the ISPOR Task Force for Translation and Cultural Adaptation. Value Health. 2005 Mar-Apr;8(2):94-104. doi: 10.1111/j.1524-4733.2005.04054.x. PMID 15804318
- [Background] Howe JA, Inness EL, Venturini A, Williams JI, Verrier MC. The Community Balance and Mobility Scale--a balance measure for individuals with traumatic brain injury. Clin Rehabil. 2006 Oct;20(10):885-95. doi: 10.1177/0269215506072183. PMID 17008340
- [Background] Inness EL, Howe JA, Niechwiej-Szwedo E, Jaglal SB, McIlroy WE, Verrier MC. Measuring Balance and Mobility after Traumatic Brain Injury: Validation of the Community Balance and Mobility Scale (CB&M). Physiother Can. 2011 Spring;63(2):199-208. doi: 10.3138/ptc.2009-45. Epub 2011 Apr 13. PMID 22379260